CLINICAL TRIAL: NCT07185087
Title: Evaluation of Treatment Progress and the Compliance of Patients Treated With DAMON Braces Versus Patients Treated With MBT Braces During Early Stage of Treatment: A Randomized Clinical Trial
Brief Title: Damon vs MBT Braces: Patient Compliance and Treatment Efficiency
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Jehan Fadhil IBrahim, Principal Investigator, Orthodontics Department, University of Baghdad, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Damon vs MBT brackets
Record Dates: First submitted 2025-08-21; First posted 2025-09-22 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Orthodontic Brackets
Keywords: Damon Ultima; Patient Compliance; MBT bracket; leveling and alignment
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Damon (Experimental): Damon Ultima Self-ligating Brackets
  Interventions: Device: passive self-ligating, Damon Ultima brackets
- MBT (Active Comparator): MBT Mini Diamond Conventional brackets
  Interventions: Device: Conventional ligation, MBT brackets

INTERVENTIONS:
Device: passive self-ligating, Damon Ultima brackets — Patients will receive Damon Ultima self-ligating brackets (Ormco Corp., Glendora, California, USA) bonded from the second molar to the second molar in each arch. Archwires will follow a standardized sequence: 0.014-inch CuNiTi, 0.018-inch CuNiTi, and 0.014 × 0.0275-inch CuNiTi (Ormco Corp., Glendora, California, USA). All bonding procedures will follow a standardized protocol, including enamel cleaning, acid etching, primer application (Ortho Solo), and adhesive curing (Green Glow).
  Arms: Damon
Device: Conventional ligation, MBT brackets — Patients will receive MBT Mini Diamond brackets (Ormco Corp., Glendora, California, USA) bonded in the same manner, with the same archwire sequence.
  Arms: MBT

SUMMARY:
Comparison between two bracket prescription systems, MBT and DAMON Ultima brackets and evaluate whether the changes incorporated in DAMON Ultima brackets can drive earlier improvement on teeth position, clinically visual progression of treatment, during initial stage of treatment. Another aim of this study is the effect of chosen bracket system on patient compliance.

DETAILED DESCRIPTION:
A single-operator, single-center randomized controlled trial (RCT) with a 1:1 allocation ratio will be conducted for patients seeking orthodontic treatment with fixed appliances. The study will take place at the Postgraduate Orthodontic Clinic, College of Dentistry, University of Baghdad, Baghdad, Iraq. Patients who meet the eligibility criteria will be randomly assigned to one of two bracket-type groups. To eliminate inter-operator variability, all patients will be treated by a single operator.

A standardized protocol will be followed. Each patient will undergo extraoral and intraoral photography, intraoral scanning with Medit i700 (Medit Corp., Seoul, South Korea), and radiographic evaluation (CBCT and lateral cephalogram). On bonding day, gingival index and plaque index will be assessed. All teeth will then be isolated and cleaned with a mixture of water and pumice using a rubber-polishing cup on a low-speed handpiece. The teeth will be rinsed and dried with an oil-free air syringe, and etched using the conventional acid-etching technique (37% orthophosphoric acid applied for 30 seconds). The surfaces will be thoroughly rinsed with water for 10 seconds to ensure complete removal of the etchant, in accordance with the manufacturer's instructions. The enamel will then be gently dried with air until a frosty-white appearance is observed.

A uniform coat of universal bonding primer (Ortho Solo, Ormco Corp., Glendora, California, USA) will be applied to the etched surfaces using a nylon bond brush. Each tooth will receive a gentle air blow for 2 seconds with the air stream directed perpendicular to the enamel surface. After etching and priming, a thin layer of adhesive (Green Glow, Ormco Corp., Glendora, California, USA) will be applied to the mesh base of each bracket, which will be positioned on the buccal surface of the tooth using a bracket holder. The bracket height will be determined according to the manufacturer's instructions. Any excess adhesive will be carefully removed from around the base of the bracket with a dental probe prior to curing, without disturbing the seated bracket. The adhesive will then be light-cured for 20 seconds.

In the intervention group, Damon Ultima brackets (Ormco Corp., Glendora, California, USA) will be bonded from the second molar to the second molar in each arch. In the comparison group, MBT Mini Diamond brackets (Ormco Corp., Glendora, California, USA) will be bonded from the second molar to the second molar in each arch. Damon Ultima archwires (Ormco Corp., Glendora, California, USA) will be used for both groups in the following sequence: 0.014-inch CuNiTi, 0.018-inch CuNiTi, and 0.014 × 0.0275-inch CuNiTi.

All patients will receive an oral hygiene kit, a brochure on dietary recommendations, and a printed questionnaire to assess pain during treatment (developed for the study). Patients will be reviewed every 8 weeks, during which gingival index, plaque index, photographs, intraoral scans, and questionnaires will be collected. Patients will also be instructed to contact the operator immediately and attend as soon as possible in the event of bracket bond failure. The treatment will be followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age range between 16-40years of age.
* ANB angle not <1° and not >5°.
* Mild to moderate crowding, spacing and rotation.
* Requiring non-extraction treatment.
* The patient agreed to be part of this study.

Exclusion Criteria:

* A history of previous orthodontic treatment with fixed appliance.
* Permanent teeth extraction except third molar.
* Congenital anomaly.
* Cleft lip and palate patients.
* Patients with ectopic canine or other teeth.
* Patients with severe crowding (<6mm).

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Degree of orthodontic treatment improvement assessed using ABO Discrepancy Index | 6 months
  Description: Evaluation of improvement in tooth rotation/alignment, overjet, overbite, occlusal relationship, interproximal contact, and cephalometric parameters.
  Time Frame: At multiple time intervals during the alignment stage (up to 6 months).
  Method: American Board of Orthodontics Discrepancy Index scoring system.
  Unit of Measure: DI points
Reduction in Malocclusion Assessed by Peer Assessment Rating (PAR) Index | 6 months
  Description: Measurement of the rate of dental alignment during treatment.
  Time Frame: At multiple time intervals during the alignment stage (up to 6 months).
  Method: Standardized PAR scoring applied to digital dental casts.
  Unit of Measure: PAR score
Improvement in Malocclusion Severity Assessed by Index of Orthodontic Treatment Need (IOTN-DHC) | 6 months
  Description: Comparison of treatment need improvement before treatment and after completion of the alignment stage.
  Time Frame: Baseline and after alignment stage (approximately 6 months).
  Method: IOTN-DHC assessment.
  Unit of Measure: IOTN grade.

SECONDARY OUTCOMES:
Changes in Oral Hygiene and Gingival Health During Treatment | 6 months
  Description: Assessment of oral hygiene and gingival health status during treatment. A composite score will be calculated by averaging Plaque Index (Silness & Löe) and Gingival Index (Löe & Silness) values.
  Time Frame: At each follow-up visit during the alignment stage (up to 6 months).
  Method: Plaque Index and Gingival Index, combined into a single composite score.
  Unit of Measure: Composite oral hygiene score.
Incidence of Bracket Bonding Failures During Treatment | 6 months
  Description: Number of bracket debonding incidents per patient during treatment.
  Time Frame: Throughout the alignment stage (up to 6 months).
  Method: Clinical records of bonding failure incidence.
  Unit of Measure: Number of debonded brackets per patient
Patient Pain Perception During Orthodontic Treatment | 6 months
  Description: Evaluation of patient pain perception during orthodontic treatment.
  Time Frame: After appliance placement and at specified time intervals during the alignment stage (up to 6 months).
  Method: Visual Analogue Scale (VAS).
  Unit of Measure: VAS score (0-10 scale).
Patient-Reported Smile Attractiveness and Confidence | 6 months
  Description: Assessment of patients' self-perception of smile aesthetics, confidence, and impact of orthodontic treatment on quality of life. Responses are collected using a structured questionnaire with multiple-choice and Likert-type questions (e.g., agreement scales, confidence levels, frequency of behaviors).
  Time Frame: Before treatment and at different time intervals during the alignment stage (up to 6 months).
  Method: Self-administered questionnaire developed for the study. Unit of Measure: Proportion of patients selecting each response category.

CONTACTS AND LOCATIONS:
Overall Officials: Jehan F. IBrahim, Principal Investigator — University of Baghdad; Hadeel A. Al-lami, Asst Prof., Study Director — University of Baghdad
Locations (1):
- University of Baghdad/ Collage of Dentistry, Baghdad, Iraq, Iraq

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD because this trial is a prospective study and yet we can't promise for any sharing

REFERENCES:
- [Background] Moyano J, Montagut D, Perera R, Fernandez-Bozal J, Puigdollers A. Comparison of changes in the dental transverse and sagittal planes between patients treated with self-ligating and with conventional brackets. Dental Press J Orthod. 2020 Jan-Feb;25(1):47-55. doi: 10.1590/2177-6709.25.1.047-055.oar. PMID 32215477
- [Background] Coenen FA, Bartz JR, Niederau C, Craveiro RB, Knaup I, Wolf M. Orthodontic treatment quality evaluated by partially automated digital IOTN and PAR index determination: a retrospective multicentre study. Eur J Orthod. 2023 May 31;45(3):308-316. doi: 10.1093/ejo/cjac064. PMID 36308300
- [Background] Barbosa IV, Ladewig VM, Almeida-Pedrin RR, Cardoso MA, Santiago Junior JF, Conti ACCF. The association between patient's compliance and age with the bonding failure of orthodontic brackets: a cross-sectional study. Prog Orthod. 2018 May 1;19(1):11. doi: 10.1186/s40510-018-0209-1. PMID 29713922
- [Background] Jahanbin A, Hasanzadeh N, Khaki S, Shafaee H. Comparison of self-ligating Damon3 and conventional MBT brackets regarding alignment efficiency and pain experience: A randomized clinical trial. J Dent Res Dent Clin Dent Prospects. 2019 Fall;13(4):281-288. doi: 10.15171/joddd.2019.043. PMID 32190212
- See also: "The Value of Self-Ligating Brackets in Orthodontics: About the Damon Protocol" (October 2021) - a chapter in Current Trends in Orthodontics by Suvetha Siva, Shreya Kishore, Suganya Dhanapal, and others — https://www.researchgate.net/publication/355885290_The_Value_of_Self-Ligating_Brackets_in_Orthodontics_About_the_Damon_Protocol